CLINICAL TRIAL: NCT00852384
Title: Non Invasive Pressure Support Ventilation (NIPPV) Versus Conventionnal Approach and Early Recruitment Maneuver (RM) for Preoxygenation of Morbidly Obese Patient
Brief Title: Non Invasive Pressure Support Ventilation (NIPPV) Versus Recruitment Maneuver (RM) and Preoxygenation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Emmanuel FUTIER, CHU Clermont-Ferrand
Allocation: Non-Randomized | Model: Parallel | Masking: Double
Other Study IDs: CHU-0046
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Obesity
Keywords: Anesthesia induction; Obese patients; Noninvasive ventilation; Alveolar recruitment
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Procedure: NIPPV and IRM — * non invasive positive pressure support ventilation (NIPPV group)
  * alveolar recruitment maneuver (IRM group)

SUMMARY:
The purpose of this study is to compare the effects of noninvasive pressure support ventilation and early alveolar recruitment maneuver during anesthesia induction of morbidly obese patients on both oxygenation and functional residual capacity modifications.

DETAILED DESCRIPTION:
Atelectasis formation during general anesthesia, leading to reduced end-expiratory lung volume, is an important cause of intrapulmonary shunt leading to impaired gas-exchange and hypoxemia. During general anesthesia and the immediate postoperative period, morbidly obese patients, who develop a larger amount of atelectasis than non-obese patient, are more likely to present impairment of gas exchange and respiratory mechanics. Noninvasive positive-pressure support ventilation (NIPPV) and positive end-expiratory pressure (PEEP) are effective to provide oxygenation during intubation of hypoxemic patients. Recent data suggest that NIPPV enhances preoxygenation in morbidly obese patients. Moreover, the application of PEEP during induction of anesthesia prevents atelectasis formation and increases nonhypoxic apnea duration in obese patients despite the use of high-inspired oxygen fraction. However, the use of both NIPPV is widely used in the operating room, because of technical and materials constraints.

Several trials have demonstrated that alveolar recruitment maneuvers (RM) are effective to remove atelectasis and improve lungs mechanics and gas-exchange.

The purpose of this randomized and controlled study is to compare the effects of two ventilatory strategies during anesthesia induction of morbidly obese patients on both gas-exchange and functional residual capacity (FRC) modifications: 1- Control group: preoxygenation using 100% O2 via a face-mask and PEEP 10 cmH2O after intubation; 2- NIPPV group: preoxygenation using NIPPV and PEEP 10 cmH2O after intubation; 3- RM group: preoxygenation using 100% O2 via a face-mask and early RM plus PEEP 10 cmH2O after intubation.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI > 30 kg/m2)
* Age > 18 years
* ASA I-III

Exclusion Criteria:

* Age < 18 years
* Patient refusal
* Pregnancy
* Emergency surgery
* COPD with FEV1 < 50%
* History of pneumothorax
* Severe asthma
* Cardiac failure (NYHA > 2)
* Ischemic heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Oxygenation (PaO2) measured 5min after the onset of mechanical ventilation | 5 min after the oneset of mechanical ventilation

SECONDARY OUTCOMES:
- FRC after tracheal intubation and after 5 min of mechanical ventilation | after 5 min of mechanichal ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Futier, Principal Investigator — University Hospital, Clermont-Ferrand; Jean-Michel Constantin, Study Director — University Hospital, Clermont-Ferrand
Locations (1):
- University Hospital Hôtel-Dieu, Clermont-Ferrand, France

REFERENCES:
- [Derived] Futier E, Constantin JM, Pelosi P, Chanques G, Massone A, Petit A, Kwiatkowski F, Bazin JE, Jaber S. Noninvasive ventilation and alveolar recruitment maneuver improve respiratory function during and after intubation of morbidly obese patients: a randomized controlled study. Anesthesiology. 2011 Jun;114(6):1354-63. doi: 10.1097/ALN.0b013e31821811ba. PMID 21478734